CLINICAL TRIAL: NCT02019576
Title: A Phase II, Multi-Centre Study, of Stereotactic Radiotherapy for Oligo-Progression in Metastatic Renal Cell Cancer Patients Receiving 1st Line Sunitinib Therapy
Brief Title: Stereotactic Radiotherapy for Metastatic Kidney Cancer Being Treated With Sunitinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZM-053
Record Dates: First submitted 2013-11-25; First posted 2013-12-24 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Clear Cell Metastatic Renal Cell Carcinoma
Keywords: Metastatic renal cell carcinoma; mRCC; Clear cell
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma; Carcinoma, Renal Cell | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: A Phase II study, single arm study, open-label, safety and efficacy study
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stereotactic radiotherapy (SRT) (Other): Stereotactic radiotherapy will be administered for up to five areas of metastatic sites showing oligo-progression within the same time period. During the Sunitinib break period, stereotactic radiotherapy will be delivered in a single fraction or up to a maximum of eight fractions. The number of fractions will depend on how many sites are being irradiated.
  Interventions: Radiation: Stereotactic radiotherapy

INTERVENTIONS:
Radiation: Stereotactic radiotherapy — SRT to all areas of oligo-progression as follows: BRAIN: 20-24 Gy in 1 fraction if < 2 cm,18 Gy in 1 fraction if 2-3 cm,15 Gy in 1 fraction for 3-4 cm, alternatively 25-30 Gy in 5 fractions can be used; SPINE: 18-24 Gy in 1-2 fractions,24 Gy in 3 fractions or 30-40 Gy in 5 fractions; NON-SPINE BONE: 30-40 Gy in 5 fractions; LUNG: 48-60 Gy in 4 fractions or 54-60 Gy in 3 fractions for peripheral lung tumours,50 Gy in 5 fractions or 60 Gy in 8 fractions for central lung tumours; LIVER: 30-60 Gy in 3-6 fractions,higher doses for central liver lesions and lower doses for peripheral liver lesions depending on proximity to adjacent organ (stomach, small bowel, large bowel or kidney); ADRENAL OR KIDNEY TUMOURS: 30-40 Gy in 5 fractions; LYMPHADENOPATHY: 30-40 Gy in 5 fractions.
  Other Names: SRT

SUMMARY:
Stereotactic radiotherapy (SRT) is a newer type of focused radiation therapy that precisely and accurately delivers high dose radiation to a tumour, while sparing much of the nearby normal organs. The use of stereotactic radiotherapy results in high rates of tumour destruction with minimal side effects which are very well tolerated. Often stereotactic radiotherapy has been used to try to cure patients who have an early stage cancer which has not spread, but there is less experience with using it in patients with cancer which has spread.

The purpose of this study is to measure how well stereotactic radiotherapy can destroy kidney cancer tumours which are no longer being controlled by Sunitinib and to measure how much longer such an approach will allow patients to stay on Sunitinib before needing to switch to another medication. Stereotactic radiotherapy will be used to treat only the growing tumours and then patients will continue with Sunitinib.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Able and willing to provide written informed consent and to comply with the study procedures.
3. Karnofsky performance status of ≥ 80%.
4. Favorable or intermediate Heng prognostic group defined as having two or less of the following factors: hemoglobin < LLN; serum corrected calcium > ULN; Karnofsky performance status < 80%; time from initial diagnosis to initiation of therapy < 1 year; absolute neutrophil count > ULN; platelet count > ULN.
5. Histologic confirmation of renal cell carcinoma with a clear cell component.
6. Evidence of measurable disease according to RECIST 1.1 criteria.
7. Already receiving first-line sunitinib therapy for at least 3 months with at least one imaging compared to baseline (or a CT from one year prior to the date of registration for patients that have been on Sunitinib therapy for over one year) that shows response or stable disease per RECIST v1.1, in all metastatic lesions (Note: SD by RECIST that allows ≤ 19% increase is allowed). Prior immunotherapy including interferon, IL-2, and checkpoint inhibitors is allowed before Sutent.
8. Radiographic evidence of ≤ 5 metastatic lesions progressing. Of the 5 progressing lesions, a maximum of 3 lesions can be in soft tissue. (Ex. If no bone metastases progressing: a maximum of 3 soft tissue lesions. If bone metastases progressing: a maximum of 5 total lesions and a maximum of 3 in soft tissue.)
9. All progressing metastases are amenable to stereotactic radiotherapy.
10. Each progression metastases fulfills at least 1 of the 3 following criteria for oligo-progression: a. Progression of an individual metastasis according to RECIST 1.1 criteria (≥ 20% enlargement of the tumour vs. baseline or nadir, taking as reference the smallest diameter seen prior to starting or during first line systemic therapy and associated with a 5 mm minimum increase in size); b. Unambiguous development of a new metastatic lesion from the time of scan taken prior to starting first-line therapy with sunitinib; c. Progressive enlargement of a known metastasis on 2 consecutive imaging studies 2-3 months apart, while receiving first-line therapy with sunitinib, with a minimum 5 mm increase in size from baseline.

Exclusion Criteria:

1. Evidence of spinal cord compression.
2. Inability to safely treat all sites of progressing metastases.
3. Prior malignancy within the past 5 years, excluding non-melanoma skin cancer and in-situ cancer.
4. Concurrent administration of other anti-cancer therapy apart from first-line sunitinib.
5. Diagnosis of ataxia telangiectasia or active collagen vascular disease.
6. Other condition, illness, psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or stereotactic radiotherapy administration, or may interfere with the interpretation of study results and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-05; Primary Completion 2021-02-16 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
To evaluate local control at one year of metastases treated with stereotactic radiotherapy in patients who present with oligo-progression while receiving first-line treatment with Sunitinib. | 3 years
  Patients will have evidence of measurable metastatic kidney cancer according to RECIST 1.1 criteria. All progressing metastases sites will be amenable to stereotactic radiotherapy. The primary endpoint of local control will be defined as the absence of local failure in the irradiated site(s). Progressive enlargement will be defined as a 20% enlargement observed on two consecutive scans from baseline scan.

SECONDARY OUTCOMES:
To evaluate progression free survival after stereotactic radiotherapy while continuing to receive first-line systemic therapy with Sunitinib. | 3 years
  Progression free survival will be evaluated via disease assessments of radiology scans completed every three months from the time of stereotactic radiotherapy until progression is confirmed. Progressive disease will be defined as a 20% increase in RECIST 1.1 criteria measurements observed on two consecutive scans from the baseline scan.
To evaluate the acute and late toxicity to stereotactic radiotherapy. | 3 years
  Acute and late toxicities to stereotactic radiotherapy will be assessed from adverse events, vital signs and by clinically significant changes in laboratory evaluations. Adverse events will use the descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. These events will be followed until resolution or for a maximum of two years, which ever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Georg A. Bjarnason, MD, FRCPC, Principal Investigator — Toronto Sunnybrook Regional Cancer Centre; Patrick Cheung, MD, FRCPC, Principal Investigator — Toronto Sunnybrook Regional Cancer Centre
Locations (12):
- Canada (12):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency, Vancouver, British Columbia
  - Manitoba CancerCare Institute, Winnipeg, Manitoba
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec